CLINICAL TRIAL: NCT06210178
Title: Non-Invasive Portal and Hepatic Vein Pressure Estimation: MRI-Guided Diagnostics for Chronic Liver Disease
Brief Title: Non-Invasive Portal and Hepatic Vein Pressure Estimation
Acronym: NONEEDLES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Hildo J Lamb, Director of Cardiovascular Imaging, Professor of Radiology, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NNDLS
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Portal Hypertension
Keywords: Magnetic Resonance Imaging; Computational Fluid Dynamics; Noninvasive; Meal challenge
MeSH Terms: conditions — Hypertension, Portal | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Other): Noninvasive MRI is performed.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — MRI scans including abdominal 4D Flow MRI.

SUMMARY:
Background Portal hypertension (PH) is a spectrum of complications of end-stage liver disease (ESLD) and cirrhosis, with severe manifestations including ascites and gastroesophageal varices. It is therefore important that timely and easily diagnosing PH has relevant prognostic and therapeutic implications. The current gold standard to evaluate PH is by hepatic vein catheterization using the transjugular approach, and measuring the hepatic venous pressure gradients (HVPG).

Time-resolved, three-dimensional, three-directional velocity-encoded MRI, also termed four-dimensional (4D) flow MRI, has been shown superior accuracy over conventional two-dimensional (2D) phase-contrast MRI, in particular for quantification of regurgitant volumes and severity of cardiac shunts. Recently, the investigators developed new imaging methods based on 4D flow MRI for visualization of the vasculature of the abdominal blood flow circulation including the portal vein. Using the newly developed computation fluid dynamics (CFD) model the investigators could determine the absolute local blood pressure in the portal vein. Preliminary data in healthy volunteers seem promising, however, data in patients with ESLD including the correlation with invasively measured HVPG are lacking.

Objectives The primary objective is to develop and validate noninvasive CFD and 4D Flow MRI based HVPG calculation to estimate portal pressure in patients with end-stage liver disease (ESLD).

Methods In 50 adult patients with ESLD, submitted for liver transplantation (LT) screening, HVPG measurements using the transjugular approach according to the standard LT screening protocol, will be extended by 4D flow MRI measurements.

Anticipated results In patients with ESLD, portal pressure can be measured by 4D flow MRI and will replace the invasive transjugular approach. The measurements can be directly incorporated in the LT screening. Moreover, the possibility to easily measure portal pressure will be relevant for all patients with ESLD at risk for PH.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will undergo a single non-invasive MRI-examination of one hour long after a four hour period of fasting. The risks associated with non-invasive MRI examinations is neglectable.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for liver transplantation (LT) screening (which excludes pregnancy).
* Age ≥ 18 years and ≤ 75 (since >75 is a contraindication for LT).
* Written informed consent.

Exclusion Criteria:

* Exclusion criteria for MRI (claustrophobia, pacemaker, metal implants, etc.).
* A psychiatric, addictive or any other disorder that compromises the subjects ability to understand the study content and to give written informed consent for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Noninvasive HVPG | Within 4 years after enrollment.
  4D Flow MRI and Computational Fluid Dynamics (CFD) based Hepatic Venous Pressure Gradient (HVPG) calculation to estimate portal pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Hildo J Lamb, PhD, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the individual participant data (IPD) outside of our research group.